CLINICAL TRIAL: NCT03009071
Title: The Effectiveness and Cost-effectiveness of Doin (Conduction Exercise) for Chronic Neck Pain: a Pilot Multicenter Randomized Controlled Clinical Trial
Brief Title: Effectiveness and Cost-effectiveness of Doin (Conduction Exercise) for Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2016-18
Record Dates: First submitted 2016-12-28; First posted 2017-01-04 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Chronic Neck Pain
Keywords: Neck Pain; Disability Evaluation; Costs and Cost Analysis; Doin Exercise Therapy; Acupuncture
MeSH Terms: conditions — Neck Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doin with Acupuncture (Experimental): An acupuncture physician will administer acupuncture at 6-12 acupoints in the upper and middle trapezius area (mandatory points: both SI15, TE15, and LI16; and selective points: GB20, BL10, GV14, SI14, and Hyeopcheok (Huatuo Jiaji, EX B2) points at C3-5 levels). Cervical Doin (conduction exercise) will be performed with the needles in situ by increasing the cervical range of motion (rotation) with physician guidance and isometric resistance exercise (rotation) as needed.
  Interventions: Procedure: Doin (conduction exercise); Device: Acupuncture
- Acupuncture (Active Comparator): An acupuncture physician will administer acupuncture at 6-12 acupoints in the upper and middle trapezius area (mandatory points: both SI15, TE15, and LI16; and selective points: GB20, BL10, GV14, SI14, and Hyeopcheok (Huatuo Jiaji, EX B2) points at C3-5 levels).
  Interventions: Device: Acupuncture

INTERVENTIONS:
Procedure: Doin (conduction exercise) — Doin (conduction exercise) will be combined with acupuncture as active and passive movement to the aim of effective treatment of pain and functional disability. Doin (conduction exercise) sessions will be conducted 2 times a week for 5 weeks.
  Other Names: Doin Exercise; Do-in Exercise; Conduction Exercise
  Arms: Doin with Acupuncture
Device: Acupuncture — Acupuncture will be performed with manual stimulation (needle twirling) to evoke de-qi sensation. Acupuncture sessions will be conducted 2 times a week for 5 weeks.

SUMMARY:
A pilot multicenter randomized controlled trial will be conducted to evaluate the clinical effectiveness, cost-effectiveness, and safety of Doin (conduction exercise) with acupuncture for chronic neck pain patients compared to acupuncture alone.

DETAILED DESCRIPTION:
A pilot multicenter randomized controlled, parallel, assessor-blinded trial will be conducted to evaluate the comparative clinical effectiveness and cost-effectiveness of Doin (conduction exercise) with acupuncture for chronic neck pain patients with acupuncture alone as assessed by pain and functional disability scales, monitor its safety, and assess the feasibility of and serve as the basis for a full-scale, multicenter trial.

ELIGIBILITY:
Inclusion Criteria:

* Onset of at least 6 months previous for neck area pain
* Current neck area pain of Numeric Rating Scale (NRS) 5 or higher
* Patients who have agreed to voluntarily participate in the clinical trial and given written informed consent

Exclusion Criteria:

* Pathologies of non-spinal or soft tissue origin or high severity which may cause neck or radiating arm pain (e.g. malignant tumor, spinal infection, inflammatory spondylitis, fibromyalgia, rheumatic arthritis, gout)
* Progressive neurologic deficit or severe neurologic symptoms (e.g. cauda equina syndrome, progressive muscle weakness)
* Other chronic diseases which may interfere with treatment effect or interpretation of results (e.g. cardiovascular disorder, renal disease, diabetic neuropathy, dementia, epilepsy)
* Current intake of steroids, immunosuppressant medicine, psychiatric medicine or other medication which may interfere with treatment results
* Patients considered unsuitable or unsafe to receive acupuncture (e.g. patients with hemorrhagic diseases, blood clotting disorders, history of anti-coagulation medicine intake, severe diabetes with high risk of infection, severe cardiovascular diseases)
* Patients who were treated with invasive interventions such as acupuncture or injections, or with medicine that may potentially influence pain such as NSAIDs (nonsteroidal antiinflammatory drugs) within the past week
* History of cervical surgery within the past 3 months
* Pregnancy or plans of pregnancy
* Severe psychopathy
* Participation in other clinical studies
* Inability to give written informed consent
* Other reasons rendering trial participation inappropriate as judged by the researchers

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Change in Northwick Park Neck Pain Questionnaire (NPQ) | 6 weeks from baseline
  Change in pain and functional disability questionnaire

SECONDARY OUTCOMES:
Northwick Park Neck Pain Questionnaire (NPQ) | Baseline (Week 1), Week 4, 6, 9, 17, 29, 53
  Pain and functional disability questionnaire
Numeric rating scale (NRS) of neck and arm pain | Baseline (Week 1), Week 2, 3, 4, 5, 6, 9, 17, 29, 53
  Pain scale
Visual analogue scale (VAS) of neck and arm pain | Baseline (Week 1), Week 2, 3, 4, 5, 6
  Pain scale
Neck Disability Index (NDI) | Baseline (Week 1), Week 4, 6, 9, 17, 29, 53
  Functional disability questionnaire
EuroQol-5 Dimension (EQ-5D) | Baseline (Week 1), Week 4, 6, 9, 17, 29, 53
  Health-related quality of life questionnaire
Patient Global Impression of Change (PGIC) | Week 4, 6, 9, 17, 29, 53
  Global, patient-reported outcome
Short Form Health Survey 12 (SF-12) | Baseline (Week 1), Week 4, 6, 9, 17, 29, 53
  Health-related quality of life questionnaire
Cost per QALY (quality-adjusted life year) | Baseline (Week 1), Week 4, 6, 9, 17, 29, 53
  Economic evaluation
Cost per NRS | Baseline (Week 1), Week 4, 6, 9, 17, 29, 53
  Economic evaluation
Drug Consumption | Baseline (Week 1), Week 2, 3, 4, 5, 6, 9, 17, 29, 53 (every visit)
  Drug type and dose of prescribe for medicine or rescue medicine, and type and frequency of other treatments (e.g. physical therapy, injection therapy)
Adverse events | Baseline (Week 1), Week 2, 3, 4, 5, 6, 9, 17, 29, 53 (every visit)
  Safety outcome

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, KMD, MPH, Principal Investigator — Jaseng Medical Foundation
Locations (1):
- Jaseng Medical Foundation, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No